CLINICAL TRIAL: NCT05993299
Title: Evaluation of Safety and Antitumor Activity of Lete-Cel (GSK3377794) in HLA-A2+ Participants With NY-ESO-1 Positive Previously Untreated Advanced (Metastatic or Unresectable) Synovial Sarcoma and Myxoid/Round Cell Liposarcoma
Brief Title: Study to Evaluate Safety and Antitumor Activity of Lete-Cel (GSK3377794) in HLA-A2+ Participants With NY-ESO-1 Positive Previously Untreated Advanced (Metastatic or Unresectable) Synovial Sarcoma and Myxoid/Round Cell Liposarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208467 Substudy 1
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-09

CONDITIONS: Neoplasms
Keywords: Adoptive T-cell therapy; Letetresgene autoleucel; Lete-cel; GSK3377794
MeSH Terms: conditions — Neoplasms | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Letetresgene autoleucel (Experimental)
  Interventions: Drug: Letetresgene autoleucel; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: Letetresgene autoleucel — Letetresgene autoleucel will be administered.
Drug: Cyclophosphamide — Cyclophosphamide will be used as a lymphodepleting chemotherapy.
Drug: Fludarabine — Fludarabine will be used as a lymphodepleting chemotherapy.

SUMMARY:
This trial will evaluate safety and efficacy of human engineered T-cell therapies, in participants with advanced tumors. This trial is a sub study of the Master study NCT03967223.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be greater than or equal to 10 years of age on the day of signing informed consent.
* Participant scheduled to receive clinical drug product supply must also weigh ≥40 kg
* Participant must be positive for HLA-A*02:01, HLA-A*02:05, and/or HLA-A*02:06 alleles by a designated central laboratory
* Participant's tumor is positive for NY-ESO-1 expression by a designated central laboratory.
* Participant has a diagnosis of synovial sarcoma (SS) or myxoid/round cell liposarcoma (MRCLS)
* Performance status: dependent on age - Lansky > 60, Karnofsky > 60, Eastern
* Cooperative Oncology Group 0-1.
* Participant must have adequate organ function and blood cell counts, within 7 days prior to leukapheresis.
* At time of treatment, participant has measurable disease according to RECIST v1.1.
* Male or female. Contraception requirements will apply at the time of leukapheresis and treatment.
* Consultation for prior history per protocol specifications.

Exclusion Criteria:

* Central nervous system metastases.
* Any other prior malignancy that is not in complete remission.
* Clinically significant systemic illness (.(Serious active infections or significant cardiac, pulmonary, hepatic or other organ dysfunction, that in the judgment of the Investigator would compromise the participant's ability to tolerate protocol therapy or significantly increase the risk of complications)
* Prior or active demyelinating disease.
* History of chronic or recurrent (within the last year prior to leukapheresis) severe autoimmune or immune mediated disease (e.g. Crohn's disease, systemic lupus) requiring steroids or other immunosuppressive treatments.
* Previous treatment with genetically engineered NY-ESO-1-specific T cells.
* Previous NY-ESO-1 vaccine or NY-ESO-1 targeting antibody.
* Prior gene therapy using an integrating vector.
* Previous allogeneic hematopoietic stem cell transplant.
* Washout periods for prior radiotherapy and systemic chemotherapy must be followed.
* Participant had major surgery in less than or equal to 28 days of first dose of study intervention.
* Prior radiation exceeds protocol specified limits.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-31 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2025-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (24):
  - City of Hope National Medical Center, Duarte, California
  - Stanford Hospital and Clinics, Stanford, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering cancer center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University-Columbus, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Hillman Cancer centre, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - University Of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (2):
  - CIUSSS de L'Est-De-Lile-De-Montreal, Montreal, Quebec
  - Princess Margaret Cancer Centre, Toronto
- France (2):
  - Centre Léon Bérard, Lyon
  - CHU de Bordeaux GH Sud Hôpital Haut Lévêque, Pessac
- Italy (2):
  - Fondazione IRCCS Instituto Nazionale Dei Tumori, Milan
  - Ircss Istituto Clinico Humanitas, Romano di Lombardia
- The Netherlands Cancer Institute, Amsterdam, Netherlands
- Spain (4):
  - Hospital Santa Creu Y Sant Pau, Barcelona
  - Ico Duran y Reynals l'Hospitalet de Llobrega, Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Virgen Del Rocio, Seville
- United Kingdom (3):
  - Royal Marsden Hospital, London
  - University College Hospital-London, London
  - Christie Hospital NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is a sub study of the master protocol (NCT03967223). The results presented are until the primary completion date. Data collection is still ongoing and additional results will be provided after study completion.
Groups:
- Letetresgene Autoleucel (Lete-cel): Eligible participants were leukapheresed to manufacture autologous lete-cel. Participants underwent lymphodepleting chemotherapy which generally consisted of fludarabine 30 mg/m^2/day on day -7 through day -4 and cyclophosphamide 900 milligrams per meter square per day (mg/m^2/day) on day -6 through day -4. followed by a single infusion of lete-cel on Day 1. The dose of lete-cel was within the range of 1×10^9 to 15×10^9 transduced T cells.
Period: Overall Study
Arm/Group | Letetresgene Autoleucel (Lete-cel)
Started | 7
Received T Cell Infusion | 5
Completed | 1
Not Completed | 6
Not completed — Did not meet treatment eligibility criteria | 2
Not completed — Ongoing | 4

BASELINE CHARACTERISTICS:
Arm/Group | Letetresgene Autoleucel (Lete-cel)
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (16.70)
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 1
  19-64 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1
  Netherlands | 2
  United Kingdom | 1
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) via investigator assessment per Response Evaluation Criteria in Solid Tumors Criteria (RECIST) version 1.1 relative to the total number of participants in the analysis population. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g., percent change from baseline). 95% CI is based on Clopper-Pearson exact confidence interval.
Time Frame: Up to approximately 36 months
Population: Modified intent-to-treat (mITT) population included all participants who received any dose of Lete-cel.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Letetresgene Autoleucel (Lete-cel)
Number analyzed (Participants) | 5
percentage of participants | 80 [28.4 to 99.5]

2. Secondary Outcome: Time to Response (TTR)
Description: Time to response was defined as the interval of time between the date of T-cell infusion and the first documented evidence of the confirmed response (PR or CR), in the subset of participants with a confirmed PR or CR as their best confirmed overall response. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g., percent change from baseline).
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2025-07

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as the interval between the initial date of confirmed response (PR/CR) and the date of progressive disease as assessed by local investigators, or death among participants with a confirmed response per RECIST 1.1. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g., percent change from baseline).
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2025-07

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with a confirmed CR, PR, or stable disease (SD) with a minimal 12 weeks (84 days ± 7 day window) duration relative to the total number of participants within the analysis population at the time of primary analysis as determined by local investigators per RECIST v1.1. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g., percent change from baseline). SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. The disease progression (PD) is defined as the date of radiological disease progression based on imaging data per RECIST v1.1. 95% CI is based on Clopper-Pearson exact confidence interval.
Time Frame: Up to approximately 36 months
Population: Modified intent-to-treat (mITT) population included all participants who received any dose of Lete-cel.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Letetresgene Autoleucel (Lete-cel)
Number analyzed (Participants) | 5
Percentage of Participants | 80.0 [28.4 to 99.5]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the interval of time between from the date of T-cell infusion to the earliest date of radiological progression of disease (PD) as assessed by local investigator per RECIST v1.1, or death due to any cause. The PD is defined as the date of radiological disease progression based on imaging data per RECIST v1.1.
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2025-07

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function.
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2025-07

7. Secondary Outcome: Number of Participants With AEs of Special Interest (AESIs)
Description: An AESI may be of scientific and medical concern related to the treatment, monitored, and rapidly communicated by investigator to sponsor. AESIs included cytokine release syndrome (CRS), hematopoietic cytopenias (including pancytopenia and aplastic anemia), graft vs host disease (GVHD), ICANS, Guillain-Barre syndrome, treatment-related inflammatory response at tumor site(s), and neutropenia Grade 4 lasting ≥28 days.
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2025-07

8. Secondary Outcome: Number of Participants With TEAEs and TESAEs by Severity
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations which involve medical or scientific judgment or is associated with liver injury and impaired liver function. AEs and SAEs were graded according to National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 5.0. Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe or medically significant but not immediately life-threatening; Grade 4- Life-threatening consequences; Grade 5- Death related to AE.
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2025-07

9. Secondary Outcome: Number of Participants With AESIs by Severity
Description: as for outcome 7
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2025-07

10. Secondary Outcome: Percentage of Participants With Replication Competent Lentivirus (RCL) Positive
Description: RCL was monitored using a polymerase chain reaction (PCR)-based assay that detects and measures copies of the gene coding for the vector's envelope protein, namely vesicular stomatitis virus G protein (VSV-G).
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2025-07

11. Secondary Outcome: Instances of Insertional Oncogenesis (IO)
Description: Instances of Insertional Oncogenesis (IO) was summarized descriptively.
Time Frame: Up to approximately 54 months
Reporting Status: Not Posted, anticipated posting 2025-07

12. Secondary Outcome: Maximum Transgene Expansion (Cmax)
Description: Cmax was defined as maximum observed persistence, determined directly from the persistence-time data. Blood samples were collected for PK analysis.
Time Frame: Day 1 to Day 14
Population: Pharmacokinetic (PK) population included participants in the safety population from whom at least one persistence sample was obtained, analyzed and was measurable.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Copies per microgram genomic DNA
Arm/Group | Letetresgene Autoleucel (Lete-cel)
Number analyzed (Participants) | 5
Copies per microgram genomic DNA | 119701.64 (68.267)

13. Secondary Outcome: Time to Cmax (Tmax)
Description: Tmax was defined as time to reach Cmax, determined directly from the persistence-time data. Blood samples were collected for PK analysis.
Time Frame: Day 1 to Day 14
Population: Pharmacokinetic (PK) population
Measure: Median (Full Range); unit: Days
Arm/Group | Letetresgene Autoleucel (Lete-cel)
Number analyzed (Participants) | 5
Days | 6.90 [1.9 to 13.6]

14. Secondary Outcome: Area Under the Time Curve From Zero to Time 28 Days (AUC[0-28])
Description: Area under the persistence-time curve from time zero to Day 28. Blood samples were collected for PK analysis.
Time Frame: Up to 28 days
Population: Pharmacokinetic (PK) population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days*copies per microgram genomic DNA
Arm/Group | Letetresgene Autoleucel (Lete-cel)
Number analyzed (Participants) | 5
Days*copies per microgram genomic DNA | 1911782.96 (53.709)

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected maximum up to approximately 36 months. Data collection is still ongoing and additional results will be provided after study completion.
Description: All-Cause mortality, Non-SAEs and SAEs were collected for intent-to-treat population that included all participants who started leukapheresis procedure.
Arm/Group | Letetresgene Autoleucel (Lete-cel)
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 4/7
Other Adverse Events (participants affected / at risk) | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letetresgene Autoleucel (Lete-cel) (N=7)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letetresgene Autoleucel (Lete-cel) (N=7)
Cytokine release syndrome (Immune system disorders) | 4 (4)
Graft versus host disease (Immune system disorders) | 1 (2)
COVID-19 (Infections and infestations) | 3 (3)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood fibrinogen decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 2 (5)
Platelet count decreased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (5)
Fatigue (General disorders) | 4 (6)
Oedema peripheral (General disorders) | 2 (2)
Axillary pain (General disorders) | 1 (1)
Catheter site phlebitis (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (4)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (3)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (2)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/99/NCT05993299/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/99/NCT05993299/SAP_001.pdf